CLINICAL TRIAL: NCT02890810
Title: Predicting Analgesic Response to Acupuncture: A Randomized, Placebo-Controlled, Subject and Assessor Blinded, 100-Subject Clinical Trial of Electro-Acupuncture in the Treatment of Chronic Low Back Pain
Brief Title: Predicting Analgesic Response to Acupuncture: A Practical Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jiang-Ti Kong, Principal Investigator, Instructor - Department of Anesthesia, Pain and Perioperative Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34754; 1K23AT008477-01A1 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-09-07 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Chronic Low Back Pain; Back Pain
Keywords: Acupuncture; Back Pain; Chronic Pain
MeSH Terms: conditions — Back Pain; Chronic Pain | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum Electroacupuncture (Experimental): Active Intervention
  Interventions: Other: Real Acupuncture with Electrical Stimulation
- Placebo Electroacupuncture (Placebo Comparator): Validated Control
  Interventions: Other: Simulated Acupuncture with Electrical Stimulation

INTERVENTIONS:
Other: Real Acupuncture with Electrical Stimulation — Acupuncture is a therapy commonly used in East Asian countries, where the practitioner insert thin needles at specific body sites in order to relieve pain and illnesses. Recent studies found low frequency electricity applied through acupuncture needles can lead to profound pain relief by increasing endorphin levels in the central nervous system. Electroacupuncture will thus be used as the active intervention to treat chronic low back pain in this clinical study.
  Other Names: Verum Electroacupuncture; Traditional acupuncture needles; ITO® ES-130® electrical stimulator
  Arms: Verum Electroacupuncture
Other: Simulated Acupuncture with Electrical Stimulation — This intervention serves as the placebo control of the active intervention. Sterile acupuncture needles and the ITO electrical stimulators will be used in this intervention. But special care will be taken to have this intervention mimic the real treatment yet remaining as physiologically inert as possible.
  Other Names: Sham Electroacupuncture / Placebo Electroacupuncture; Sterile Acupuncture Needles; ITO® ES-130® electrical stimulator
  Arms: Placebo Electroacupuncture

SUMMARY:
In this placebo controlled, patient and assessor blinded clinical trial, the investigators will administer electroacupuncture vs sham electroacupuncture to patients suffering from chronic low back pain, and monitor their symptoms as well as collecting objective outcome measures. The investigators objective is to identify predictors of pain reduction and functional improvement with electroacupuncture vs placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65
2. English Fluency
3. Chronic LBP for ≥ 6 Months

   1. Chronicity: cLBP "defined as a back pain problem that has persisted at least 3 months and has resulted in pain on at least half the days in the past 6 months."
   2. Location: "between the lower posterior margin of the rib cage and the horizontal gluteal fold
4. Average pain over the last month ≥ 5/10

Exclusion Criteria:

1. Radicular low back pain: defined as sharp (or burning) pain, with a defined territory, radiating down the limb, beyond the knee. Radicular pain may be accompanied by sensory and motor deficit along 1 or more dermatomes. Radicular back pain may also be accompanied by MRI evidence of intervertebral disc protrusion and compression of spinal cord and/or nerve roots.
2. Pending litigation or Worker's compensation related to the low back pain.
3. Currently pregnant or planning to become pregnant (in next 6 months)
4. American Society of Anesthesiologist (ASA) class III or above physical status. ASA class III is defined as "a patient with severe systemic disease." Examples would include poorly controlled diabetes, hypertension, COPD or morbid obesity (BMI ≥ 40).
5. Mental health conditions or treatment for mental health problems that would interfere with study procedures, at the discretion of the study team. For example, psychosis, untreated major depression, ongoing substance abuse, suicidal ideation. These will be assessed by the MINI.
6. Medications: opioids ≥60mg morphine equivalent units/day, benzodiazepines, corticosteroids.
7. Prohibited interventions: during the study period, the following are not permitted

   1. Back surgeries
   2. Injections with local anesthetics or steroids to the back
   3. New chiropractic maneuvers
   4. New physical therapy programs
   5. New medications for back pain
8. Bleeding disorders at the discretion of the study team.
9. Previous acupuncture treatment in the past 10 years.
10. Medical conditions that would interfere with study procedures (eg. Heart disease or pacemaker, active infection), per discretion of the team

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Mean back pain intensity by patient-report | 7 days
  Patient self-reported mean back pain intensity on 11 point (0-10) numerical rating scale (NRS).
Roland Morris Disability Questionnaire | 1 day
  Validated functional outcome measure in chronic low back pain with 24 yes/no questions regarding physical function.

SECONDARY OUTCOMES:
Quantitative Sensory Testing | Tests used are typically stable for 1-2 weeks
  Standardized response to noxious thermal and mechanical stimuli up to 120 seconds.
Physical exam to determine neurological function | 1 month
  Physical exam assessing neurological function (recorded as presence or absence of light touch sensation, and stretch reflexes at the knees and ankles) in up to 5min.
Physical exam to assess lumbar facet irritation. | 1 month
  Physical exam assessing facet irritation via positive or negative response to lumbar facet maneuver in up to 5 minutes.
Physical exam to assess lumbar spine range of motion | 1 month
  Physical exam assessing range of motion in lumbar spine (measured in degrees) in up to 5 minutes.
Blood pressure | 1 day
  Blood pressure collected via OMRON electric blood pressure monitor, in mmHg up to 60 seconds.
Heart Rate Variability | 1 month
  Heart rate variability (LF/HF) collected via non-invasive, HRVLive! device up to 10 minutes.
Heart Rate Variability | 1 month
  Heart rate variability (BPM) collected via non-invasive, HRVLive! device up to 10 minutes.
Heart Rate Variability | 1 month
  Heart rate variability (ECG) collected via non-invasive, HRVLive! device up to 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Systems Neuroscience and Pain Lab (SNAPL), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kong JT, Puetz C, Tian L, Haynes I, Lee E, Stafford RS, Manber R, Mackey S. Effect of Electroacupuncture vs Sham Treatment on Change in Pain Severity Among Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2022787. doi: 10.1001/jamanetworkopen.2020.22787. PMID 33107921